CLINICAL TRIAL: NCT02924324
Title: RePPAIR -Reducing Procedural Pain and Improving Recovery of Quality of Life in Pediatric Neuroblastoma Patients Undergoing Bone Marrow Procedures: A Prospective Randomized Cross-over Clinical Trial
Brief Title: Local Injection of Pain Medication to Reduce Pain After Bone Marrow Procedures in Pediatric Neuroblastoma Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 16-1417
Record Dates: First submitted 2016-10-03; First posted 2016-10-05 (Estimated); Results first posted 2022-04-26 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2021-10

CONDITIONS: Neuroblastoma
Keywords: local Injection; pain Medication; propofol; ropivacaine; 16-1417
MeSH Terms: conditions — Neuroblastoma | interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Propofol First, then Propofol & Ropivacaine (Active Comparator): 1st Bone Marrow procedure (BM) Intervention A: propofol first. Then second BM procedure with propofol & ropivacaine
  Interventions: Device: propofol; Behavioral: Wong-Baker FACES® Pain Rating Scale; Behavioral: Post-procedural quality of life (QOL)
- Propofol and Ropivacaine First, then Propofol (Experimental): 1st BM procedure: Intervention B: propofol & ropivacaine first. Then second BM procedure with propofol
  Interventions: Drug: ropivacaine; Behavioral: Wong-Baker FACES® Pain Rating Scale; Behavioral: Post-procedural quality of life (QOL)

INTERVENTIONS:
Device: propofol
  Arms: Propofol First, then Propofol & Ropivacaine
Drug: ropivacaine
  Arms: Propofol and Ropivacaine First, then Propofol
Behavioral: Wong-Baker FACES® Pain Rating Scale — Nurses will record patient-reported pain scores.
Behavioral: Post-procedural quality of life (QOL)

SUMMARY:
The purpose of this study is to identify whether or not the addition of a numbing medicine that is injected directly into the site of the bone marrow procedure can reduce pain and the use of opioid pain medication after bone marrow procedures. The addition of this medicine, called ropivacaine, is the experimental part of this study. This is the first time ropivacaine will be directly injected into the bone marrow site at MSKCC Pediatrics.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of neuroblastoma as defined by the International Neuroblastoma Risk Group Staging System (INRGSS)22
* 3 - 18 years of age
* Patient has had prior bone marrow procedures
* English speaking

Exclusion Criteria:

* History of allergy to investigational agent: ropivacaine or other amino amide analgesics
* History of allergy to standard agent: propofol
* Chronic daily opioid requirement
* Lansky/Karnofsky Score < 60
* Inability to comply with protocol requirements including refusal to forego pre-procedural opioid use
* Patient is receiving additional potentially painful interventions (e.g. central line insertion/removal) concurrent with the bone marrow procedure

Ages: 3 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 56 (Actual)
Dates: Start 2016-10; Primary Completion 2019-11 (Actual); Study Completion 2019-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ellen Basu, MD, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center, New York, New York, United States

REFERENCES:
- [Derived] Zarnegar-Lumley S, Lange KR, Mathias MD, Nakajima-Hatano M, Offer KM, Ogu UO, Ortiz MV, Tan KS, Kellick M, Modak S, Roberts SS, Basu EM, Dingeman RS. Local Anesthesia With General Anesthesia for Pediatric Bone Marrow Procedures. Pediatrics. 2019 Aug;144(2):e20183829. doi: 10.1542/peds.2018-3829. PMID 31366683
- See also: Memorial Sloan Kettering Cancer Center — https://www.mskcc.org/

RESULTS

PARTICIPANT FLOW:
Groups:
- Propofol With Placebo First Then Propofol With Ropivacaine: ARM 1: 1st Bone Marrow procedure (BM) Intervention A: propofol first. Then second BM procedure with propofol & ropivacaine
- Propofol With Ropivacaine First Then Propofol With Placebo: ARM 2: 1st BM procedure: Intervention B: propofol & ropivacaine first. Then second BM procedure with propofol
Period: Overall Study
Arm/Group | Propofol With Placebo First Then Propofol With Ropivacaine | Propofol With Ropivacaine First Then Propofol With Placebo
Started | 28 | 28
Completed | 28 | 28
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Propofol With Placebo First Then Propofol With Ropivacaine | Propofol With Ropivacaine First Then Propofol With Placebo | Total
Number analyzed (Participants) | 28 | 28 | 56
Age, Continuous [Median (Full Range); unit: years] | 7.75 [3 to 16] | 6.5 [3 to 14] | 7.13 [3 to 16]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 7 | 20
  Male | 15 | 21 | 36
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 28 | 27 | 55
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 1 | 3 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 3 | 4
  White | 23 | 19 | 42
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 2 | 5
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 28 | 27 | 55
  United Kingdom | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Requiring Post-procedural Opioid Analgesia Per Study Arm
Description: Number of participants requiring post-procedural opioid analgesia within 24 hours (+/- 4 hours) post procedure per study arm
Time Frame: within 24 hours (+/- 4 hours) post procedure
Measure: Number; unit: participants
Groups:
- Propofol Alone: Participants who received propofol alone
- Propofol & Ropivacaine: Participants who received propofol & ropivacaine
Arm/Group | Propofol Alone | Propofol & Ropivacaine
Number analyzed (Participants) | 56 | 56
participants
  Require postprocedural opioid | 22 | 22
  Did not Require postprocedural opioid | 34 | 34

ADVERSE EVENTS:
Time Frame: Up to 1 year
Groups:
- Propofol: Participants received propofol alone
- Propofol and Ropivacaine: Participants received propofol & ropivacaine in combination
Arm/Group | Propofol | Propofol and Ropivacaine
All-Cause Mortality (participants affected / at risk) | 12/56 | 12/56
Serious Adverse Events (participants affected / at risk) | 0/56 | 0/56
Other Adverse Events (participants affected / at risk) | 0/56 | 0/56

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-01-30): https://cdn.clinicaltrials.gov/large-docs/24/NCT02924324/Prot_SAP_000.pdf